CLINICAL TRIAL: NCT04861922
Title: Low Dose Unfractioned Heparin for Treatment of Sepsis Caused by Abdominal Infection：a Pilot Study
Brief Title: Unfractioned Heparin for Treatment of Sepsis Caused by Abdominal Infection
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Collaborators: Xiangya Hospital of Central South University (Other); Central South University (Other); The Second Hospital University of South China (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); The Affiliated Yantai Yuhuangding Hospital of Qingdao University (Unknown)
Responsible Party: Principal Investigator, Ben Lu, Principal Investigator, The Third Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XY3-UFH2021
Record Dates: First submitted 2021-04-22; First posted 2021-04-27 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Sepsis; Gram-Negative Bacterial Infections; Heparin
MeSH Terms: conditions — Sepsis; Gram-Negative Bacterial Infections | interventions — Heparin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unfractionated Heparin (Experimental): A bottle solution of Heparin Sodium (2ml:12500IU) is added to 48 ml saline and administered intravenously continuously for 24 hours (10 unit/kgBW/hour), which last 5 days or until the death or discharge.
  Interventions: Drug: Unfractionated Heparin
- Normal saline (Placebo Comparator): The same amount of 0.9% saline as the heparin group (50ml) will be administered in the placebo group.
  Interventions: Drug: Unfractionated Heparin

INTERVENTIONS:
Drug: Unfractionated Heparin — 10 unit/kgBW/hour continuous infusion for 5 days
  Other Names: Heparin sodium

SUMMARY:
Sepsis is the leading cause of death in intensive care units and a major public health concern in the world. Heparin, a widely used anticoagulant medicine to prevent or treat thrombotic disorders, has been demonstrated to prevent organ damage and lethality in experimental sepsis models. However, the efficacy of heparin in the treatment of clinical sepsis is not consistent. Caspase-11, a cytosolic receptor of LPS, triggers lethal immune responses in sepsis. Recently, we have revealed that heparin prevents cytosolic delivery of LPS and caspase-11 activation in sepsis through inhibiting the heparanase-mediated glycocalyx degradation and the HMGB1- LPS interaction, which is independent of its anticoagulant properties. In our study, it is found that heparin treatment could prevent lethal responses in endotoxemia or Gram-negative sepsis, while caspase-11 deficiency or heparin treatment failed to confer protection against sepsis caused by Staphylococcus aureus, a type of Gram-positive bacterium. It is probably that other pathogens such as Gram-positive bacteria might cause death through mechanisms distinct from that of Gram-negative bacteria. Peptidoglycan, a cell-wall component of Gram-positive bacteria, can cause DIC and impair survival in primates by activating both extrinsic and intrinsic coagulation pathways, which might not be targeted by heparin. We speculate that the discrepancy between the previous clinical trials of heparin might be due to the difference in infected pathogens. Thus, stratification of patients based on the type of invading pathogens might improve the therapeutic efficiency of heparin in sepsis, and this merits future investigations.

DETAILED DESCRIPTION:
In clinical patients, the major pathogens of sepsis caused by abdominal infection are mostly Gram-negative bacterium. Therefore, aim of this study is to determine effects of low dose unfractionated heparin for treatment of sepsis caused by abdominal infection.

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible for inclusion if all of the inclusion criteria are met:

1.Sepsis-3 criteria from Society of Critical Care Medicine (SCCM) /European Society of Intensive Care Medicine (ESICM), and the infection site is from abdomen 2.18≤ age ≤75years 3.obtain informed consent

Exclusion Criteria:

1. The primary site of infection is from other parts (such as lungs, intracranial, etc.) except abdomen
2. Diagnosis of sepsis for more than 48 hour
3. Pregnant and lactating women
4. Severe primary disease including unrespectable tumours, blood diseases and Human Immunodeficiency Virus (HIV);
5. Have a known or suspected adverse reaction to UFH including HIT
6. Have bleeding or high risk for bleeding
7. Have an indication for therapeutic anticoagulation or have taken anticoagulants within 7 days
8. Use of an immunosuppressant or having an organ transplant within the previous 6 months
9. Participating in other clinical trials in the previous 30 days
10. Have received cardiopulmonary resuscitation within 7 days
11. Have terminal illness with a life expectancy of less than 28 days

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-05-11 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
All-Cause Mortality | 28 Days after randomization
  Death from all causes at 28-days

SECONDARY OUTCOMES:
Death in ICU | 28 Days after randomization
  Death from all causes at ICU discharge
SOFA score | Day 0,3,6 after randomization
  Total Sequential Organ Failure Assessment (SOFA) score(0-24) , higher values represent a worse outcome
APACHEⅡ | Day 0,3,6 after randomization
  Acute Physiology and Chronic Health Evaluation (include Acute physiology score, APS and age and Chronic physiology score, totally 0-71 Points)
SIC score | Day 0,3,6 after randomization
  Sepsis-induced coagulopathy score (totally 0-6 Points)
DIC score | Day 0,3,6 after randomization
  Disseminated intravascular coagulation score (totally 0-8 Points)
Duration of mechanical ventilation and continuous renal replacement therapy | 28 days after randomization
  Duration of mechanical ventilation and continuous renal replacement therapy in ICU
ICU stay | 28 days after randomization
  Duration of stay in ICU
Inflammation | 0,3,6 days after randomization
  Concentration of inflammation markers such as c-reactive protein, procalcitonin, IL-1β and IL-1α at 0, 3,6 days after randomization
Coagulation | 0,3,6 days after randomization
  Concentration of coagulation related indexes such as fibrinogen degradation products, d-dimer, thrombin-antithrombin complex, plasminogen activator inhibitor-1, plasmin antiplasmin complex, and thrombomodulin at 0,3,6 days after randomization
The incidence of major bleeding | 28 days after randomization
  "Major bleeding" is defined as intracranial bleeding, life-threatening bleeding, or need red blood cell suspension more than 3 units every 24 hours, and last for 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Hong Yuan, MD, Study Chair — The third Xiangya Hospital, Central South University
Locations (1):
- The third Xiangya Hospital, Central South University, Changsha, Hunan, China

REFERENCES:
- [Background] Tang Y, Wang X, Li Z, He Z, Yang X, Cheng X, Peng Y, Xue Q, Bai Y, Zhang R, Zhao K, Liang F, Xiao X, Andersson U, Wang H, Billiar TR, Lu B. Heparin prevents caspase-11-dependent septic lethality independent of anticoagulant properties. Immunity. 2021 Mar 9;54(3):454-467.e6. doi: 10.1016/j.immuni.2021.01.007. Epub 2021 Feb 8. PMID 33561388
- [Background] Deng M, Tang Y, Li W, Wang X, Zhang R, Zhang X, Zhao X, Liu J, Tang C, Liu Z, Huang Y, Peng H, Xiao L, Tang D, Scott MJ, Wang Q, Liu J, Xiao X, Watkins S, Li J, Yang H, Wang H, Chen F, Tracey KJ, Billiar TR, Lu B. The Endotoxin Delivery Protein HMGB1 Mediates Caspase-11-Dependent Lethality in Sepsis. Immunity. 2018 Oct 16;49(4):740-753.e7. doi: 10.1016/j.immuni.2018.08.016. Epub 2018 Oct 9. PMID 30314759
- [Background] Yang X, Cheng X, Tang Y, Qiu X, Wang Y, Kang H, Wu J, Wang Z, Liu Y, Chen F, Xiao X, Mackman N, Billiar TR, Han J, Lu B. Bacterial Endotoxin Activates the Coagulation Cascade through Gasdermin D-Dependent Phosphatidylserine Exposure. Immunity. 2019 Dec 17;51(6):983-996.e6. doi: 10.1016/j.immuni.2019.11.005. Epub 2019 Dec 10. PMID 31836429
- [Background] Yang X, Cheng X, Tang Y, Qiu X, Wang Z, Fu G, Wu J, Kang H, Wang J, Wang H, Chen F, Xiao X, Billiar TR, Lu B. The role of type 1 interferons in coagulation induced by gram-negative bacteria. Blood. 2020 Apr 2;135(14):1087-1100. doi: 10.1182/blood.2019002282. PMID 32016282
- [Background] Lu Y, Meng R, Wang X, Xu Y, Tang Y, Wu J, Xue Q, Yu S, Duan M, Shan D, Wang Q, Wang H, Billiar TR, Xiao X, Chen F, Lu B. Caspase-11 signaling enhances graft-versus-host disease. Nat Commun. 2019 Sep 6;10(1):4044. doi: 10.1038/s41467-019-11895-2. PMID 31492850